CLINICAL TRIAL: NCT06461299
Title: A Single-Center Pilot Study to Evaluate the Efficacy, Safety, and Tolerability of Sarecycline for Treating Periorificial Dermatitis
Brief Title: Study to Evaluate the Efficacy, Safety, and Tolerability of Sarecycline for Treating Periorificial Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Dermatology Institute of Boston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIB-0601
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Perioral Dermatitis
MeSH Terms: conditions — Dermatitis, Perioral

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, pilot study to evaluate the efficacy, safety, and tolerability of sarecycline (Seysara) for periorificial dermatitis. This will be a four-week open-label study using sarecycline to treat POD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- A Single-ARM Pilot Study to Evaluate Sarecycline for Treating Periorificial Dermatitis (Experimental): A Single-Center Pilot Study to Evaluate the Efficacy, Safety, and Tolerability of Sarecycline for Treating Periorificial Dermatitis
  Interventions: Drug: Seysara Oral Product

INTERVENTIONS:
Drug: Seysara Oral Product — Subjects with a clinical diagnosis of POD will be given sarecycline for four weeks. Dosing of sarecycline will be weight based, either 60mg, 100mg, or 150mg PO qday. Each subject will have at least three visits, including a screening/baseline visit, a two-week follow-up, and a four-week follow-up. The initial diagnosis will be made by a board-certified dermatologist or a dermatology-certified nurse practitioner. The Perioral Dermatitis Severity Index, PODSI, (Appendix I) will be used to grade the severity of periorificial dermatitis throughout the three visits. This published scoring method ranges from 0 to 9. To be included in the study, patients must need to have a PODSI score of "moderate" (PODSI = 3.0-5.5) or "severe" (PODSI = 6.0-9.0) at baseline. The primary endpoint is the percentage of patients that receive a PODSI score ranging from 0 ("none") to 2.5 ("mild") at week four. The secondary endpoint is the patient reported an adverse event at week four.

SUMMARY:
A Single-Center Pilot Study to Evaluate the Efficacy, Safety, and Tolerability of Sarecycline for Treating Periorificial Dermatitis

DETAILED DESCRIPTION:
This pilot study's intended purpose is to evaluate the efficacy, safety, and tolerability of sarecycline for periorificial dermatitis. Sarecycline, a third-generation tetracycline, is currently only indicated to treat acne vulgaris. However, the investigator has used sarecycline to treat periorificial dermatitis and would like to capture and report on this efficacy in a pilot study. The investigator hypothesize's that not only will the subjects respond well to sarecycline treatment, but that it will be well-tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of POD by both the principal investigator and a blinded observer
* Have a PODSI score of 3.0 or greater at baseline by clinical investigator
* Must not be dysphagic.
* Patient is male or female, 18-55 years of age inclusive at Screening.

Exclusion Criteria:

* Allergy to tetracyclines.
* Immunocompromised.
* Pregnancy or planning a pregnancy during the study period.
* Lactating subjects.
* Ongoing use of any of the following treatments to the face throughout study; oral or topical steroids, oral or topical calcineurin inhibitors, topical retinoids, topical antibiotics, - oral or topical metronidazole, or topical azelaic acid.
* Facial hair or skin dermatoses that interfere with evaluation of the perioral dermatitis.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
PODSI score | 4 weeks
  The PODSI represents the sum of individual scores for erythema, papules and scaling. Each of these key features is graded on a scale from 0 to 3 including intermediate values (0.5, 1.5 and 2.5). The PODSI is defined as the sum score of the 3 features, and may range from 0 to 9. All patients with a PODSI from 0.5 to 2.5 were regarded as mild, whereas severe cases scored with a PODSI from 6.0 to 9.0. All remaining patients with a PODSI from 3.0 to 5.5 were classified as moderate.

CONTACTS AND LOCATIONS:
Locations (1):
- The Dermatology Institute of Boston, Boston, Massachusetts, United States